CLINICAL TRIAL: NCT04761315
Title: Detecting Atrial Fibrillation in Patients With an Embolic Stroke of Undetermined Source (From the DAF-ESUS Registry)
Status: Completed | Type: Observational
Sponsor: Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other)
Responsible Party: Sponsor
Other Study IDs: TFM 2016-18
Record Dates: First submitted 2020-11-11; First posted 2021-02-18 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Fibrillation, Atrial
Keywords: cardiac implantable electronic devices; interatrial block; P-wave duration
MeSH Terms: conditions — Atrial Fibrillation; Interatrial Block

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The presence of interatrial block (IAB) is associated with the development of atrial fibrillation (AF). The aim of this study was to determine whether P-wave duration and presence of IAB before the implantation of a cardiac implantable electronic device (CIED) are associated with the presence of atrial high rate episodes (AHRE), during long-term follow-up.

DETAILED DESCRIPTION:
The presence of interatrial block (IAB) is associated with the development of atrial fibrillation (AF). The aim of this study was to determine whether P-wave duration and presence of IAB before the implantation of a cardiac implantable electronic device (CIED) are associated with the presence of atrial high rate episodes (AHRE), during long-term follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients in sinus rhythm
* with or without previous paroxysmal AF
* with dual-chamber pacemakers (PMs), implantable cardioverterdefibrillators (ICDs), and devices for cardiac resynchronization therapy (CRT)
* capable of atrial activity monitoring were included in the study

Exclusion Criteria:

-Previous documented atrial fibrillation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in sinus rhythm, with or without previous paroxysmal AF and with dual-chamber pacemakers (PMs), implantable cardioverterdefibrillators (ICDs), and devices for cardiac resynchronization therapy (CRT) capable of atrial activity monitoring were included in the study
Sampling Method: Non-Probability Sample
Enrollment: 380 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Atrial high rate new episodes | 24 months
  New episodes of atrial high rate episodes